CLINICAL TRIAL: NCT03299634
Title: Prevalence of Oral Mucosal Lesions Among Smokers in an Egyptian Cohort: A Hospital-based Cross-Sectional Study (I)
Brief Title: Oral Mucosal Lesions Among Smokers in an Egyptian Population Study.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amira Mohamed Abdel-aziz, resident, Cairo University
Other Study IDs: CEBC-CU-2017-08-05
Record Dates: First submitted 2017-09-28; First posted 2017-10-03 (Actual); Last update posted 2017-10-20 (Actual); Status verified 2017-10

CONDITIONS: Smokers

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Histopathological evaluation of clinically suspicious oral lesions to detect dysplasia (Warnakulasuriy et al., 2007 and Rastogi et al., 2013).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: printed questionnaire — For each eligible participant, a full history will be obtained according to a questionnaire followed by thorough clinical examination.

SUMMARY:
This cross-sectional study will assess the prevalence of oral changes among smokers in an Egyptian cohort (patients attending to the hospital of Faculty of Dentistry - Cairo University), aiming that this study can serve as a baseline for future studies with the goal of finding ways to improve oral health and increase awareness of the hazards of smoking in Egypt

DETAILED DESCRIPTION:
The participants will be selected from the pool of the Clinics of Oral Medicine, Periodontology and Diagnosis Department and the Diagnostic center, Faculty of Dentistry - Cairo University. For each eligible participant, a full history will be obtained according to a questionnaire followed by thorough clinical examination.

ELIGIBILITY:
Inclusion Criteria:

* Gender: males and females.
* Age: all age groups.
* Smokers.
* Individuals who agreed to sign the informed consent.

Exclusion Criteria:

* Individuals suffering from any systemic disease.
* Individuals on medications.
* Non-Egyptians.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The participants will be selected from the pool of the Clinics of Oral Medicine, Periodontology and Diagnosis Department and the Diagnostic center, Faculty of Dentistry - Cairo University. For each eligible participant, a full history will be obtained according to a questionnaire followed by thorough clinical examination.
Sampling Method: Probability Sample
Enrollment: 840 (Estimated)
Dates: Start 2017-11-01 (Estimated); Primary Completion 2018-11-30 (Estimated); Study Completion 2018-12-01 (Estimated)

PRIMARY OUTCOMES:
oral mucosal lesions | one year
  Identifying and recording oral mucosal lesions

SECONDARY OUTCOMES:
Oral health-related quality of life (OH-QoL) evaluation | one year
  using Oral Health Impact Profile (OHIP)
dysplasia | one year
  Histopathological evaluation of clinically suspicious oral lesions to detect dysplasia